CLINICAL TRIAL: NCT04164537
Title: Patient, Family, and Provider Perspectives on Latina Adolescents' Depression Treatment Engagement
Brief Title: Latina Adolescent Depression Treatment Study
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00103001; U54MD012530 (NIH)
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Depression
Keywords: Hispanic Americans, Adolescent
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Latina adolescents and parents: Latina adolescent young women experiencing depression and their parents will be recruited from community and primary care settings for one-time individual interviews.
- Healthcare providers: Primary care and mental health providers who commonly work with Latina adolescent patients will be recruited for focus groups from an integrated primary care clinic.

SUMMARY:
Despite experiencing higher rates of depressive symptoms and similar rates of Major Depressive Disorder (MDD), Latina (female) adolescents in the U.S. are significantly less likely than their non-Latina White peers to receive treatment for MDD. The purpose of this study is to identify facilitators of and barriers to depression treatment engagement among Latina adolescents across patient-, family-, and healthcare provider-levels from the perspectives of these individuals. Latina adolescent-parent dyads and healthcare providers will be recruited from community and healthcare settings. Separate individual semi-structured interviews will be conducted with Latina adolescents (n=12) and their parents (n=12). Two focus groups will be conducted with primary care providers (n=6) and mental health providers (n=6) who frequently care for Latina youth. Qualitative content analysis will be used to analyze the transcripts to determine common themes in facilitators and barriers across stakeholder groups.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* Ages 13-17
* Self-identify as Hispanic/Latina
* Be first generation (i.e. born outside the US) or second generation immigrants (i.e. one or both parents born outside the US)
* Have been diagnosed with Major Depressive Disorder or Persistent Depressive Disorder/Dysthymia
* Have been referred to psychotherapy or prescribed medication for depression

Adolescent Exclusion Criteria:

* Currently experiencing acute psychological distress

Parent Inclusion Criteria

* Parent of Latina adolescent experiencing depression

Parent Exclusion Criteria

* Not fluent in English or Spanish

Healthcare Provider Inclusion Criteria

* Self-identify as regularly providing clinical care to Latina adolescents with depression
* Be in a role in which they can refer to or provide depression treatment

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Patient self-report of female gender identity.
Study Population: Latina adolescent young women experiencing depression and their parents will be recruited from community and integrated primary care settings. Healthcare providers will be recruited from an integrated primary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of barriers to depression treatment among Latina adolescents generated from patient interviews and provider focus groups | Baseline
Number of facilitators of depression treatment among Latina adolescents generated from patient interviews and provider focus groups | Baseline
Number of preferences for depression treatment generated from patient interviews and provider focus groups | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Gonzalez-Guarda, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Lincoln Community Health Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No